CLINICAL TRIAL: NCT06755840
Title: Sleep Disordered Breathing and Multimorbidity: The Xiangya SDB Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024080978
Record Dates: First submitted 2024-11-21; First posted 2025-01-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disordered Breathing (SDB); Sleep Apnea; Cardiometabolic Diseases; Multimorbidity; Neurodegenerative Diseases
Keywords: sleep disordered breathing; obstructive sleep apnea; central sleep apnea; cardiovascular diseases; metabolic diseases; respiratory diseases; nervous system diseases; mental disorders; neoplasms; multimorbidity
MeSH Terms: conditions — Sleep Apnea Syndromes; Neurodegenerative Diseases; Sleep Apnea, Obstructive; Sleep Apnea, Central; Cardiovascular Diseases; Metabolic Diseases; Respiratory Tract Diseases; Nervous System Diseases; Mental Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep disordered breathing (SDB) is one of the most common sleep disorders, including obstructive sleep apnea (OSA), central sleep apnea (CSA), sleep-related hypoventilation, hypoxemia, etc., with OSA being the most prevalent. Also, SDB shows high comorbidities with multisystem diseases. Furthermore, compared to patients with pure SDB, those comorbid with SDB and other disorders like cardiometabolic dysfunction and cognitive impairment experience poorer quality of life, higher rate of disease progression and mortality, and a greater economic burden. Currently, there are limited cohorts to study the associations between SDB and multisystem diseases. The aim of this study is to establish an ambispective clinical cohort for SDB in Xiangya hospital from central-south China (Xiangya Sleep Disordered Breathing Cohort, Xiangya SDB cohort) including retrospective part and prospective part, which covers multi-dimensional data of sleep monitoring, demographic, daily behaviors, clinical manifestations and comorbidities status, life quality, treatment information and evaluation, etc. by self-reported questionnaires and objective assessments and tests. Besides, whole peripheral blood is drawn for following biomarkers study and omics analysis. The main goal is to achieve precise management of SDB and related multimorbidity, containing to early identify risk individuals for multisystem impairment, significantly improve their prognosis and ultimately enhance overall health. In detail: first, to reveal how multisystem impairment related to SDB evolves; second, to identify which indicators closely involve system dysfunction due to SDB; third, to build an efficient model and a cost-effective platform to screen high-risk population and tract therapeutic effect.

DETAILED DESCRIPTION:
This study will be designed as a non-interventional and ambispective cohort study incorporating a retrospective part (Xiangya SDB cohort-Retrospective part) and a prospective part (Xiangya SDB cohort-Prospective part). It has received approval from the Medical Ethics Committee of Xiangya Hospital Central South University on August 21, 2024. The study will collect basic information, sleep parameters, clinical manifestation, comorbidities status, life quality and mortality from participants, through subjective and objective questionnaires, physical examinations, sleep monitoring, laboratory tests (blood routine test, serum biochemistry, myocardial enzymes, etc.), imaging tests (CT, echocardiogram, etc.) and other specific tests (pulmonary function test, etc.), as well as subsequent annual visits.

Xiangya SDB cohort-Retrospective part: The participants in this part primarily include individuals who completed sleep monitoring at the Sleep Medicine Center of Xiangya Hospital of Central South University from January 1, 2016 to January 14, 2025. Relevant comorbidities diagnoses and treatment data will be extracted from electronic health records. Meanwhile, questionnaires, physical examinations, laboratory tests, imaging tests, echocardiograms and pulmonary function tests, etc. will also be accessed to evaluate multisystem function and impairments. Subsequent long-term visits will collect all-cause and specific-cause death and evaluate the improvement and/or progression of cardiovascular, metabolic, respiratory, nervous, mental and neoplastic disorders, with supplementary data gathered from historical records.

Xiangya SDB cohort-Prospective part: The prospective cohort will begin enrolling participants from January 15, 2025, with their first sleep monitoring and the date of enrollment as the baseline visit. Concurrently, their basic information, clinical data, questionnaires related to sleep habits and quality, comorbidities status, physical examination, hospital laboratory and imaging data and pulmonary function test, etc. will also be collected. Subsequently, participants will be followed up every 12 to 24 months through phone calls, home visits or hospital visits.

Notably, participants signing informed consent will have an additional 10 ml of peripheral blood collected during routine clinical care (outpatient visits, hospitalizations, follow-ups, etc.) for biomarkers and multi-omics research. The follow-up visits will include: 1) death event and the causes; 2) relevant questionnaires and tests described as above to assess the function and diseases disease status of each comorbid system.

ELIGIBILITY:
Inclusion Criteria:

* 1) Participants who were suspected of sleep disordered breathing must complete at least one overnight sleep monitoring at the Sleep Medicine Center at Xiangya Hospital.
* 2) Participants can finish any assessment for each comorbid system by questionnaires, scales, physical examinations and tests, etc. independently or with the assistance.
* 3) Participants agreed to participate in this study with signing an informed consent form.

Exclusion Criteria:

* Participants who refused to participate in this study or whose clinical data was lost.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: participants who complete at least one overnight sleep monitor session in the Sleep Medicine Center of Xiangya hospital Central South University
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-10-31 (Estimated)

PRIMARY OUTCOMES:
Death event | From participants agreed to participate in this study until the date of death from any or specific cause or the end of the study, whichever came first, assessed up to 10 years.
  Death due to any cause or specific cause

SECONDARY OUTCOMES:
Life quality as measured by the 12-item short form health survey (SF-12) | Through study completion, an average of 2 years
  The seven situations of SF-12 include physical function, role limitations due to physical health or emotional problems, bodily pain, general health perceptions, vitality, and social function. The scoring criteria for the SF-12 scale is based on a percentage system, where higher scores indicate better quality of life.
Daytime sleepiness as measured by the Epworth Sleepiness Scale (ESS) | Through study completion, an average of 2 years
  ESS is intended to assess sleepiness liability (from 0 to 3 score) across eight different situations, the higher score indicates more likely to sleepiness.
Sleep quality and behavior as measured by the Pittsburgh Sleep Quality Index (PSQI) | Through study completion, an average of 2 years
  The seven different dimensions of PSQI include sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The total score of PSQI ranges from 0 to 21 and the higher score indicates poorer sleep.
Rapid Eye Movement Sleep Behavior Disorder Questionnaire Hong Kong (RBD-HK) applied for RBD screening | Through study completion, an average of 2 years
  RBD-HK mainly accesses symptoms and severity of RBD.
Cognitive function and impairment as measured by Ascertain Dementia 8 (AD8) | Through study completion, an average of 2 years
  AD8 is intended to access cognitive function and impairment through eight concise questions. A score of 2 or above indicates cognitive impairment.
Number of participants with cardiometabolic diseases or events | Through study completion, an average of 2 years
  The occurrence of cardiometabolic diseases or events (e.g. hypertension, heart failure, ACS and DM, etc.) are identified by self-report or their electronic health records and tests (e.g. blood pressure, blood glucose, lipids and hormone levels, echocardiogram, ECG etc.)
Number of participants with respiratory diseases or events | Through study completion, an average of 2 years
  The occurrence of respiratory diseases or events (e.g. COPD and asthma, or hospitalization due to exacerbation, etc.) are identified by self-report or their electronic health records and tests (e.g. lung function test parameters, etc.)
Number of participants with nervous system and mental diseases and status | Through study completion, an average of 2 years
  The occurrence of nervous system and mental diseases and status (e.g. stroke, dementia, Parkinson's disease, depression, etc.) are identified by participants self-report or their electronic health records.
Number of participants with digestive system diseases or events | Through study completion, an average of 2 years
  The occurrence of digestive diseases (e.g. GERD, crohn's disease, ulcerative colitis, etc.) are identified by participants self-report or their electronic health records
Number of participants with kidney diseases or events | Through study completion, an average of 2 years
  The occurrence of kidney diseases or events (e.g. CKD etc.) are identified by self-report or their electronic health records and tests (e.g. eGFR etc.)
Number of participants with neoplasms diseases or events | Through study completion, an average of 2 years
  The occurrence of neoplasms diseases or events (e.g. any type of tumor, adverse events, etc. ) are identified by self-report or their electronic health records

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No